CLINICAL TRIAL: NCT02995538
Title: Neurogenetics Program Patient Registry: Clinical and Genetic Diagnosis, Natural History Study, Translational Research and Biorepository
Brief Title: Neurogenetics Patient Registry
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Deepa Soundara Rajan, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY19090278
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Neurogenetic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Biospecimen Retention: Samples With DNA — Blood samples and tissue samples if available after completion of tests ordered on these patients for clinical purposes will be de-identified and stored to create a biorepository. DNA sample from genetic testing that is left over after appropriate clinical testing will be used for storage at the biorepository and for further appropriate research testing.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Neurogenetic Patients: The Neurogenetics Clinic, which started in 2016, provides clinical care for undiagnosed patients with complex neurological disorders in which a genetic etiology is considered and for children with diagnosed rare neurogenetic disorders - provide pre test counseling, diagnostic services for the undiagnosed patients and long-term management of patients with a wide range of diagnosed genetic disorders of the nervous system.

SUMMARY:
The objective of this project is to develop a Neurogenetics patient database and bio repository - which includes clinical information regarding history, physical examination, laboratory testing including genetic testing (NextGen sequencing including whole exome and whole genome sequencing, SNParray, etc.), neuroradiology studies, neurophysiology studies - all ordered as clinically deemed appropriate, natural history from clinical longitudinal follow-up and to use de-identified information from this registry/ repository, when appropriate for clinical and translational research.

DETAILED DESCRIPTION:
Patients seen in the neurogenetics clinic with a clinical phenotype or a pedigree supportive of a genetic disease will be considered for the study. Autosomal recessive inheritance will be suggested by at least two affected sibs with healthy parents who may also have other unaffected children. Autosomal dominant inheritance will be suggested by multiple affected family members in multiple generations. Lack of family history could be suggestive of autosomal recessive inheritance or de novo autosomal dominant inheritance.

Informed consent will be completed prior to any research procedures or genetic testing. Patients seen in the neurogenetics clinic will be approached about participating in the Neurogenetics study during their routine clinic visit. Parents of pediatric patients seen in the clinic will be asked to provide their written informed consent. Following informed consent, deidentified patient information will be entered in a database by a study team member. If participation in the biorepository is also approved, then available stored specimens will be deidentified and located in the specific laboratories or in a collaborators laboratory

In the case of a known Neurogenetics patient who has died, the Legally Authorized Representative (or next of kin) of a deceased patient may be approached to provide permission for research data and stored specimens to be included in this study. Again, their protected health information (including any samples that were clinically obtained from biopsies or at autopsy) will be secured and de-identified for their participation.

Immediate family members will be studied (affected individual, affected and unaffected siblings and parents) with the goal of studying at least a family in trio (mother, father, affected child). In some cases, the family may have a deceased individual with banked DNA available. If the family is interested in including these samples, written consent will be obtained from the decedent's next-of-kin or the executors of the decedent' estate.

Family history suggestive of genetic disease which is undiagnosed with the available diagnosis methods will be considered for the study after having an extensive genetic evaluation. Affected individuals beside their affected and unaffected siblings and both their parents will be considered for the study.

The research subjects will be seen by a member of the study team to discuss the research protocol and obtain informed consent. They will also be seen in the clinic once we have the final results of the research study for genetic counseling and to discuss the results. If needed they will be seen in the clinic for other clinical reasons that are not related to the research.

Methodology:

For Goal 1: A neurogenetics clinic has been set up with 2 clinical child neurologists and a genetic counselor, where undiagnosed patients with a potential neurogenetic disease will be assessed and clinically appropriate testing will be ordered. Patients with diagnosed neurogenetic disorders will also be followed for longitudinal care and reassessment as appropriate.

For Goal 2: Informed consent will be obtained and pretesting genetic counseling will be provided. Clinically appropriate testing will be ordered including blood draw, urine specimen collection, buccal swab collection and if needed tissue biopsy samples. DNA sample from the above testing that is left over after appropriate clinical testing will be used for storage at the biorepository and for further appropriate research testing. Next generation sequencing, if clinically appropriate will be ordered through available commercial labs as approved by the patient's insurance company. If insurance coverage is denied research testing will be ordered after informed consent and pretesting counseling, to be done through our collaborative labs.

For Goal 3: A patient database with de-identified clinical information, laboratory analysis, imaging studies and genetic studies will be maintained. A biorepository of blood and other DNA/ tissue samples will be maintained in the appropriate clinical / collaborators laboratory. The patient database will facilitate and identification and recruitment of potential eligible subjects for the participation in patient specific translational research studies to help better delineate the patients condition or to help with potential therapy development in the future.

Collaborators have been identified in multiple different fields through the university of Pittsburgh to help with offering research next generation testing, bioinformatics analysis, basic science researchers to help with functional analysis of potential novel genes/ variants of unknown significance. The vision of the initiative is to be able to take data from novel new genetic testing on undiagnosed patients to the bench for functional characterization - with the hope that this would pave the road to repurposing currently available drugs for personalized care of these rare patients or help development of novel treatments in the future.

Experimental Approach:

Blood draw will be ordered as clinically indicated with an extra tube been drawn for research purposes: Up to 20 mL of whole blood will be collected in EDTA tubes. DNA will be extracted per standard lab protocols. For deceased individuals we will be using banked source of DNA if available. Next of kin will sign proxy consent for deceased individuals. Whole Exome Sequencing (exome amplification and sequencing) and/or Whole Genome Sequencing will be done according to lab protocol and will be sent out to a commercial laboratory or a laboratory in consultation with one of our collaborators/consultants on this protocol. Research whole exome through a collaborators laboratory will be offered to patients, whose insurance providers will not cover for clinical testing.

The bioinformatics analysis provided by collaborators will be used to analyze the raw data from NGS. Standard analysis will be used looking for variants in specific genes known to cause genetic disorders. Any variants on whole exome or whole genome sequencing found will then be compared to publicly available exomes/genomes from the dbSNP database, 1000 Genome Project and NHLBI (http://evs.gs.washington.edu/EVS/) to exclude common variants and will be compared to data available from ClinVar (http://www.ncbi.nlm.nih.gov/clinvar/) as well as ExAC (ExAC.broadinstitute.org). Variants pathogenic prediction using available software such as PolyPhen and SIFT will be used in the analysis as well. Comparing variants found in an affected individual to those found in each parent further reduces the number of candidate variants. For autosomal dominant disorders, this strategy can discover de novo coding variants, assuming neither parent is a non-expressing carrier of the disorder. In contrast, in recessive disorders each parent should carry one of the disease-causing variants identified in the affected children. For X- linked disorders, the mother should be carrier for the disease unless it has occurred de novo in the proband. Conservation score such as GERP score (Genomic Evolutionary Rate Profiling) will be noted as well. Alteration of a highly conserved residue is more likely to be functionally significant. Genes with multiple transcripts will require special consideration. In this situation, effect estimation will be limited to those from canonical transcripts, variants in candidate genes will then be confirmed by Sanger sequencing in a CLIA certified lab.

Assessment of Physiologic Relevance: Based on published literature reports of similar experiments, we anticipate that we will identify <10 candidate genes and perhaps as few as one. If more than one candidate gene is identified, we will assess likely physiologic relevance a number of ways. First, amino acid changes will be assessed for conservation across evolution. Alteration of a highly conserved residue is more likely to be functionally significant. Next we will assess predicted tissue expression through examination of EST databases and "virtual northern blots". Amino acid changes predicted to significantly alter protein structure will be assessed further by doing functional studies.

Time Frame and Subsequent Studies: The proposed sequencing studies can be completed relatively expediently once sample is obtained. Additional time will be required for bioinformatic analysis. Data obtained through this project will be used by the PI to prepare grant applications to systematically characterize the underlying molecular defects in patients with significant pedigree evidence of a genetic disorder, or in patients with recognized genetic syndromes of unknown cause. Preliminary data obtained through this project will also lead to additional grant applications to study the identified defect.

The blood draw will be done on the affected individuals, healthy parents and unaffected siblings in the phlebotomy lab at Children's Hospital of UPMC or other UPMC facilities where patients are seen by the lab personnel. The blood draw should take no more than 5-10 minutes. Alternate arrangements may be made with individuals and their local phlebotomy lab to obtain the specimens and ship them to the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patients evaluated at the Neurogenetics clinic and suspected to have an underlying neurogenetic disorder will be included.
* Patients with known abnormal genetic testing with a neurological phenotype will be included.

Exclusion Criteria:

* Patient with acquired diagnosis, which can explain the patients clinical symptoms and with a clinical phenotype or family history not suggestive of an underlying genetic etiology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neurogenetics Patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Genetic testing | Within approximately one year for each participant
  Next generation sequencing, if clinically appropriate will be ordered through available commercial labs as approved by the patient's insurance company. If insurance coverage is denied research testing will be ordered after informed consent and pretesting counseling, to be done through our collaborative labs.

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Soundara Rajan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Results relevant to the participant's clinical condition will be verified in a CLIA-certified laboratory and reported to the participant.